CLINICAL TRIAL: NCT00150839
Title: Hippocampal Volume in Young Patients With Major Depression Before and After Combined Antidepressive Therapy - a Monocentric, Double-blind, Placebo-controlled Trial
Brief Title: Hippocampal Volume in Young Patients With Major Depression Before and After Combined Antidepressive Therapy
Acronym: COATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Stefan Bleich, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COATS
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Venlafaxine; Mirtazapine; Double-blind RCT; Magnetic resonance imaging; Hippocampal volume
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mirtazapine; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Probands receive mirtazapine and venlafaxine
  Interventions: Drug: Venlafaxine
- 2 (Placebo Comparator): Patients receive mirtazapine and placebo
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Mirtazapine — Patients receive mirtazapine 45mg and placebo.
  Other Names: Remergil SolTab (R)
  Arms: 2
Drug: Venlafaxine — Patients receive mirtazapine 45mg and venlafaxine 300mg.
  Other Names: Remergil SolTab (R); Trevilor retard (R)
  Arms: 1

SUMMARY:
The proposed study is a randomized, placebo-controlled, double-blind trial to evaluate the safety and efficacy of antidepressant combination for the treatment of depression.

Depressive disorder is one of the most common human diseases with a high burden for every patient, her/his family, health care system and society as a whole. Actual treatment concepts of depressive disorders include pharmacologic, biologic (e.g. electroconvulsive therapy, light therapy) and psychologic therapy. Even though effective therapeutic options are at hand, therapy needs time. It is often not possible to reach full remission of the disease and 10-25% of patients suffering from depression are regarded as "treatment-resistant". In treatment resistant depression, the use of a combination of antidepressive drugs is considered safe and effective. However, at present no data exist concerning the use of drug combination as primary therapeutic option. The aim of the study is to examine the hypothesis, that significantly more patients achieve full remission of depressive symptoms when treated with the combination of two antidepressants and as a secondary hypothesis, that patients receiving a drug combination will achieve remission faster than patients treated with monotherapy. To test these hypotheses, a two group parallel design is used comparing the efficacy and safety of mirtazapine in combination with venlafaxine or placebo.

DETAILED DESCRIPTION:
Background Information

Combining antidepressants is a well-established medical procedure for the treatment of therapy refractory depression, that may also be applied successfully under non-refractory conditions. The goal of the study is to test this hypothesis. All participants are to be treated with Remergil Soltab®, a sedative antidepressant containing mirtazapine. In a double-blind, parallel-group design, all participants are treated with either Trevilor® retard, an antidepressant of the selective-serotonin-norepinephrine-reuptake-inhibitor class containing venlafaxine or placebo.

Especially in the treatment of therapy-resistant depression augmentation- and combination strategies are widely used (Demling and Frieling 2004).

Only limited data exist on the efficacy and safety of combination of antidepressants: Carpenter et al. have shown, that adjunctive use of mirtazapine added to the prior used antidepressant (mostly SSRIs) was more effective than placebo (Carpenter et al 2002). Devarajan and Dursun report a more effective antidepressive therapy with the combination of citalopram and reboxetine (Devarajan and Dursun 2000). Rubio et al. found the combination of reboxetine, SSRI or venlafaxine and mirtazapine effective (Rubio et al 2004). Smith et al. report less side effects of venlafaxine use when combined with mirtazapine.

All mentioned studies were conducted in treatment-resistant depression. Only the study by Carpenter et al. was done in a randomized, controlled, double-blind design. No data exist on the efficacy and safety of combined antidepressant use as primary therapy of depression.

Pallanti et al. were able to show, that combination of SSRI and mirtazapine leads to an earlier onset of therapeutic effects in OCD (Pallanti et al 2004).

There exists little evidence on the benefits of combined antidepressant use in depression. However, combination of antidepressants proved to be effective and safe in treatment-resistant depression. All used antidepressants have side-effects (see "Fachinformation" for further details). Drug-drug interactions have not been described for the drugs used in the trial. A risk-potentiation therefore seems unlikely.

Route of administration:

Venlafaxine and placebo are administered orally, the usual mode of administration for antidepressive drugs. Only Remergil Soltab®is administered using an orodispersible tablet. This way of administering mirtazapine has proven to be effective.

Dosage:

All participants are to be treated with Remergil Soltab® 45mg, the highest dosage of its license in Germany.

Trevilor® retard will be used 300mg/d. It is licensed for 375mg/d, but for practicability reasons, especially blinding procedures, the modestly lower dosage will be entertained.

Dosage regimen:

Remergil® medication starts with 15mg for two days after randomization. On day 3 and 4, 30mg are used. From day 5 on, 45mg are used.

In the Trevilor® group, treatment starts with 150mg for the first three days, afterwards 300mg are used.

Beginning with day 4, both groups are treated with two capsules of the blinded study medication.

Treatment period:

All patients are treated for 12 weeks in a double-blind fashion.

The trial will be conducted in compliance with this protocol, the guidelines for good clinical practice (CPMP/ICH/135/95) and the applicable regulatory requirements, namely the German law on drugs (AMG).

Participants:

160 participants, both female and male are to be recruited when admitted to the open wards of the Department of Psychiatry and Psychotherapy, Universitätsklinikum Erlangen. Participants have to suffer from depressive disorder and need to be 18-65 years old.

Treatment of Subjects

After screening and inclusion into the trial, all prior psychopharmacological medication is stopped and washed out. How dose reduction and cessation is done will be decided individually. The wash-out phase should not exceed 5-7 days. The use of irreversible inhibitors of monoamine oxidase (MAOI) during 14 days prior to screening is an exclusion criterion, as a wash-out period of 14 days is not suitable for the trial. After the wash-out, patients are randomized into two groups:

1. VENLA - Participants receiving Trevilor®retard 150mg in a blinded capsule. For three days, one capsule is administered, afterwards two capsules are administered, representing a dosage of 300mg/d.
2. CONT - Participants receiving placebo capsules. For three days, one capsule is administered, afterwards two capsules are administered.

All participants are receiving Remergil Soltab® starting with 15mg for two days, 30mg for days 3 and 4 and 45mg beginning with day 5

Medication permitted during the trial: all non-psychiatric medication, lorazepam and pipamperon.

Medication not permitted: Antidepressants other than the study medication, neuroleptics other than pipamperon, sedative other than lorazepam. Medication with known interactions with the study medication (according to the SPC).

All medication is allowed before the wash-out period of the trial with the exception of irreversible MAO inhibitors (MAOI).

Medication permitted after the trial: All medication is allowed after the trial. The use of MAOI and other monoaminergic substances should not be started earlier than 14 days after the end of intake of study medication.

Assessment of Efficacy

Efficacy is assessed using different psychometric scales either filled out by the participant or the investigator. Scales to be used are BDI, BAI, BSI, PSQuI as questionaires filled by the participant and CGI, MADR-S, HAM-D and HAM-A as rating scales filled out by the investigator. During the first week and week 13, a cranial magnetic resonance image is obtained, to assess morphologic changes of the brain.

During the weekly visits, BDI, BAI, CGI, HAM-D, HAM-A and MADR-S are entertained. BSI and PSQuI are entertained at screening, visit 4, visit 8, visit 12 and visit 13. (please see also the attached flow chart and 16 Supplement A for further details).

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18-55 years
* Moderate to severe depressive episode according to ICD10-criteria ICD10:F32.1, F32.2, F33.1, F33.2) and MADRS-sum value >=18 points

Exclusion Criteria:

* Bipolar affective disorder incl. BD-II.
* Psychiatric or neurologic comorbidity.
* Depression with psychotic symptoms.
* Pregnancy or lactation period.
* Significant cardiovascular or gastrointestinal disease.
* Severe dysfunction of liver (defined according to Child-Pugh-Criteria (>=Child A)) or kidney (defined according to KDIGO stage I (albuminuria >=30mg/g).
* Known and proven pharmacoresistance.
* Proven contraindication against MRI (e.g. pacemaker).
* Known incompatibility against one of the substances used.
* Intake of irreversible inhibitors of monoamine oxidase (MAOI, e.g. tranylcypromine) during last 14 days.
* Known phenylketonuria.
* Women with childbearing potential not using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Categorial response to the medication. Categorial response is defined on the basis of CGI Improvement scale and 50% reduction in MADR-S score | Whole duration of study

SECONDARY OUTCOMES:
Tolerability of treatment as assessed using the DOTES scale | Whole duration of study
Cognitive deficits as judged by the SKT system | Study duration
Self assessment of depression and anxiety using Beck's Depression/Anxiety Inventory (BDI/BAI) | Whole study
Changes is blood levels of homocysteine, folate, vit B12, P11 | whole study duration

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bleich, MD, Principal Investigator — University Erlangen-Nuremberg
Locations (1):
- Department of Psychiatry and Psychotherapy, University Erlangen-Nuremberg, Erlangen, Bavaria, Germany